CLINICAL TRIAL: NCT03973853
Title: The Importance of the Nurse's Role in Treatment Observance and Social Autonomy in Schizophrenia Using an Innovating Tool for Daily Transports: a Pilot Study
Brief Title: How Can a Driving Virtual Reality Tool Improve Quality of Life and Social Autonomy in Patients With Schizophrenia
Acronym: Schizovirt
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision to stop the study
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-A02799-46
Record Dates: First submitted 2019-04-25; First posted 2019-06-04 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
Keywords: virtual reality; social autonomy; road safety; driving abilities; schizophrenia; cognitive functioning
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group with virtual reality stimulation (Experimental): The subjects in this arm will undertake 14 sessions of virtual reality stimulation. The program will be delivered by a nurse, trained to the use of such a tool, and familiar with cognitive remediation techniques. Before and after these 14 sessions, social autonomy, daily life skills, cognitive domains and self-esteem will be measured
  Interventions: Behavioral: Virtual reality driving stimulation program
- Treatment as Usual group (TAU) (Placebo Comparator): Patients in this group will carry on benefiting from their usual care with no additional program. They will be assessed before and after a 3 month period for social autonomy, daily life skills, cognitive domains and self-esteem.
  Interventions: Behavioral: TAU

INTERVENTIONS:
Behavioral: Virtual reality driving stimulation program — This group will benefit of 14 one hour sessions, using the driving simulator. The program is based on a progressive training, focused on the remediation of the cognitive functions specific to driving. The tool and the type of training aim to help transfer the abilities to daily life.
  Arms: Active group with virtual reality stimulation
Behavioral: TAU — This group will carry on their usual treatment during the whole length of the study. Patients will be randomized into the 2 groups. This TAU group will be the control group and will help assess the effectiveness of the stimulation program. The stimulation sessions will be proposed to the TAU group at the end of study.
  Arms: Treatment as Usual group (TAU)

SUMMARY:
Schizophrenia is a mental health issue that affects mostly young adults. The main symptoms are hallucinations, delirium, and agitation, poor social relations, lack of motivation, thought disorganization. Also, patients suffering from schizophrenia encounter important cognitive disorders affecting memory, executive functioning and attention. These cognitive alterations are often linked to social exclusion and stigmatisation.

Antipsychotic treatments are effective mainly on the positive dimension of symptoms (hallucinations etc…); however their action is very limited on the cognitive difficulties encountered. Psychosocial techniques can be used to treat the cognitive symptoms, such as cognitive remediation or psychosocial rehabilitation .

These cognitive difficulties mainly have an impact on patients' daily life, affecting their abilities to drive, for example. Schizophrenic patients suffer more road accidents than healthy subjects .

Thus, considering this information, it appears important to us to address this driving problem for various reasons:

* Firstly, knowing how to drive is often linked to daily autonomy,
* Secondly, driving is also linked to keeping an active social network and to work.

Patients suffering from schizophrenia often encounter difficulties in learning how to drive which reinforces the stigmatisation and fear of failure.

Thus, a specific driving and theory training prior to driving lessons could be a way of helping patients in their cognitive difficulties and pass their driving test. Daily transports mobilize a number of cognitive functions (attentional vigilance, working memory, psychomotor coordination, divided attention, visuo-spatial abilities .

Using a driving virtual reality tool could constitute an ecological cognitive remediation tool, by simulating daily driving situations. This "serious game" approach enables us to involve virtual reality in training but also in assessments. The driving simulator allows standardized evaluations and could also become a therapeutic tool of ecological cognitive remediation.

This study thus appears interesting in order to develop road safety and daily autonomy.

DETAILED DESCRIPTION:
In order to study the impact of a driving virtual reality tool on daily autonomy and cognitive functioning, patients will undertake a number of training sessions using the tool.

This study will be composed of 2 groups of schizophrenic patients.

* the active group will benefit from 14 one hour sessions on the driving simulator. The training will be progressive and organized enabling the remediation of the different cognitive functions necessary to driving.
* the TAU (treatment as usual) group will carry on their usual care during the length of the study. This group will help confirm the pertinence of using such a tool on a daily basis. After the end of the study, the 14 session training will be suggested to the patients who are willing.

Social autonomy, neuropsychological functioning and clinical symptomatology will be measured before, after and at a 6 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic of Schizophrenia according to a DSM-5 criteria
* Aged between 18-50 years
* Enrolled in an empowerment project
* Stable clinical status, without treatment modification for 3 months
* Capacity to consent
* Affiliated to a social security scheme

Exclusion Criteria:

* Opposition of patient or legal guardian
* Background of head trauma, neurological pathology with cerebral repercussions or severe somatic or ocular disease not stabilized or resulting in pain> 3 months
* Visual disorders related to surgery or known ocular pathology leading to visual loss or visual field restriction
* Mental retardation < 80
* Simultaneous participation in another cognitive remediation program (6-month exclusion period)
* Simultaneous participation in another study involving cognitive processes (6-month exclusion period)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Social Autonomy | 7 months
  the primary outcome will be the modification before and after intervention of the total score on the Social Autonomy scale. It is obtained by 5 domains (personal health, everyday life, money, social relationships, and affective life).

SECONDARY OUTCOMES:
Rosenberg Self-esteem | 7 months
  the outcome measure of self esteem will be the modification before and after the score of scale. It is a brief auto-questionnaire.
World Health Organization Quality of Life Assessment (WHOQLOL-BREF) | 7 months
  the quality of life will be evaluated before and after intervention
The positive and negative syndrome (PANSS) | 7 months
  the measure of cognitive functioning specific to the driving situation will be the modification before and after intervention of the score obtained at the proposed neuropsychological evaluation (executive, attentional and social)
Car Simulator Evaluation Test | 7 months
  Change in score "Car Simulator Evaluation Test" . This measure is repeated at the beginning and at the end of the intervention to highlight the impact of the " Car Simulator " program, and 6 months later to investigate the benefits.
  the impact of the program on road safety knowledge outcome will be assessed by the modification before and after of scores using the assessments available with the driving tool

CONTACTS AND LOCATIONS:
Overall Officials: ROMAIN REY, PH, Principal Investigator — CH Le Vinatier
Locations (2):
- France (2):
  - Hôpital le vinatier, Bron
  - Hopital Vinatier, Bron